CLINICAL TRIAL: NCT03542669
Title: A Phase I Study of Autologous Killer Cell Injection Induced by Dendritic Dells Loaded With 6B11 Anti-idiotype Minibody (6b11 - OCIK Injection) Treatment in Patients With Recurrent Drug-resistant Ovarian Cancer
Brief Title: Study of 6b11-OCIK Injection Treatment in Patients With Recurrent Drug-resistant Ovarian Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Weixiao Biotechnology Development Limited (Industry)
Responsible Party: Principal Investigator, Changxiaohong, Director of Gynaecologic Oncology Center, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6B11-OCIK-I
Record Dates: First submitted 2018-05-20; First posted 2018-05-31 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Recurrent Ovarian Carcinoma; Platinum-resistant Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6B11-OCIK injection (Experimental)
  Interventions: Drug: 6B11-OCIK Injection; Drug: Doxorubicin

INTERVENTIONS:
Drug: 6B11-OCIK Injection — Two infusions of 6B11-OCIK will be performed at each chemotherapy cycle (Day 3 an Day 7) during the first three cycles, while PBMC will be collected before each cycle (Day -12) during the first three cycles.
Drug: Doxorubicin — Subjects will be adminitered 4~6 cycles of chemotherapy (Doxorubicin, 30 mg/m^2 IV on Day 1 of every cycle)

SUMMARY:
This is an open, single-arm, phase I clinical trial to evaluate safety and efficacy and of 6b11-OCIK injection in the treatment of recurrent drug-resistant ovarian cancer

DETAILED DESCRIPTION:
This is a phase I clinical trial of cytotoxic T cell injection induced by dendritic cells loaded with 6B11 anti-idiotype minibody (6b11-OCIK injection) for recurrent drug-resistant ovarian cancer. Main purpose of this research is to determine the maximum tolerable dose (MTD) of 6B11-OCIK injection in the treatment of patients with ovarian cancer. Moreover, secondary purpose is to evaluate the effect of 6B11-OCIK injection on the immune system of patients, the efficacy of autologous 6B11-OCIK injection in the treatment of patients with ovarian cancer obtain and the correlation between OC166-9 antigen expression and efficacy of 6B11-OCIK injection. Thirdly, exploratory purpose is to evaluate the effect of 6B11-OCIK injection on laboratory examination.

ELIGIBILITY:
Inclusion criteria:

1. 18-70 years old patients.
2. Diagnosed as Ovarian Cancer, who had relapsed after initial treatment; Relapse after drug resistance: clinical remission after early chemotherapy, but progression or relapse within 6 months after chemotherapy,or achieve no response after early chemotherapy.
3. Administered with Doxorubicin.

Exclusion criteria:

1. Symptomatic and uncontrolled Brain metastasis or pia meningeal metastasis; Patients with spinal cord compression; Symptoms related to central nervous system lesions or symptoms indicating disease progression;
2. Corticosteroid drugs (or analogues) or drugs effecting the immune system were administered before infusion in 4 weeks.
3. Patients with interstitial lung disease or interstitial pneumonia, including clinically significant radiation pneumonia;
4. Women with positive serum pregnancy test or lactation;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2018-08-03 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
MTD | 1 year
  Determine the maximum tolerable dose (MTD) of 6B11-OCIK injection in the treatment of patients with ovarian cancer base on the AE, SAE and laboratory examination.

SECONDARY OUTCOMES:
Changes of the cell immunophenotype | 1 year
  Changes in the concentrations of the cell immunophenotype (CD3+, CD3+CD4+, CD3+CD8+, CD3-CD56+, CD3-CD19+) in peripheral blood after 6B11-OCIK injection from baseline.
Changes of the antinuclear antibody (ANA) | 1 year
  Changes in the concentrations of the antinuclear antibody (ANA) in peripheral blood after 6B11-OCIK injection from baseline.
Changes of the C-reactive protein (CRP) | 1 year
  Changes in the concentrations of the C-reactive protein (CRP) in peripheral blood after 6B11-OCIK injection from baseline.
Changes of the interleukin-6 (IL-6) | 1 year
  Changes in the concentrations of the interleukin-6 (IL-6) in peripheral blood after 6B11-OCIK injection from baseline.
Changes of the immunoglobulin | 1 year
  Changes in the concentrations of the immunoglobulin in peripheral blood after 6B11-OCIK injection from baseline.
Objective response rate (ORR) | 3 years
  Percentage of patients who achieved CR and PR after treatment.
Disease control rate (DCR) | 3 years
  Percentage of evaluable patients who achieved CR, PR and SD after treatment.
Progression Free Survival (PFS) | 3 years
  The period from the first infusion of 6B11-OCIK to first PD or death from any cause.
Correlation between OC166-9 antigen expression and efficacy of 6B11-OCIK injection. | 1 year
  OC166-9 antigen expression and efficacy of 6B11-OCIK

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohong Chang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng H, Ma R, Wang S, Wang Y, Li Y, Tang Z, Dou S, Wang Y, Zhu H, Ye X, Zhang T, Zhang Y, Li S, Zhao Y, Li Y, Cui H, Chang X. Preliminary Safety and Potential Effect of 6B11-OCIK Adoptive Cell Therapy Against Platinum-Resistant Recurrent or Refractory Ovarian Cancer. Front Immunol. 2021 Aug 2;12:707468. doi: 10.3389/fimmu.2021.707468. eCollection 2021. PMID 34408750
- See also: Preliminary Safety and Potential Effect of 6B11-OCIK Adoptive Cell Therapy Against PlatinumResistant Recurrent or Refractory Ovarian Cancer,Frontiers in immunology,2021,12:707468 — http://doi.org/10.3389/fimmu.2021.707468